CLINICAL TRIAL: NCT03691454
Title: A Randomized, Multicenter, Controlled, Adaptive II/III Study to Compare Neoadjuvant Chemotherapy of Docetaxel，Oxaliplatin Combined With S-1(DOS) Versus Oxaliplatin Combined With S-1(SOX)in Locally Advanced Gastric Adenocarcinoma (RESOLVE-2 Study)
Brief Title: Compare Neoadjuvant Chemotherapy of DOS Versus SOX in Locally Advanced Gastric Adenocarcinoma.
Acronym: RESOLVE-2
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Head of Beijing Cancer Hospital, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGOG1008
Record Dates: First submitted 2018-09-11; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Gastric Adenocarcinoma
Keywords: gastric adenocarcinoma; neoadjuvant chemotherapy; locally advanced; Oxaliplatin; S-1; Docetaxel
MeSH Terms: interventions — Docetaxel; Oxaliplatin; S 1 (combination); Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DOS (Experimental): Docetaxel+Oxaliplatin+S-1
  Interventions: Drug: Docetaxel
- SOX (Active Comparator): Oxaliplatin+S-1
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 50mg/m2, intravenous drip, D1, combined with Oxaliplatin 85mg/m2，intravenous drip 2h，D1 and S-1 40-60mg bid(BSA<1.25m2, 40mg bid, 1.25m2≤BSA≤1.5m2, 50mg bid, BSA>1.5m2, 60mg bid)，D1-7；For patients with Her2 positive, add Herceptin 4mg/kg(6mg/kg first cycle) D1; every 14 days for a cycle.
  Other Names: Oxaliplatin; S-1; Herceptin
  Arms: DOS
Drug: Oxaliplatin — Oxaliplatin 130mg/m2，intravenous drip 2h，D1 combined with S-1 40-60mg bid(BSA<1.25m2, 40mg bid, 1.25m2≤BSA≤1.5m2, 50mg bid, BSA>1.5m2, 60mg bid)，D1-14；For patients with Her2 positive, add Herceptin 6mg/kg(8mg/kg first cycle) D1; every 21 days for a cycle.
  Other Names: S-1; Herceptin
  Arms: SOX

SUMMARY:
This is a randomized, multicenter, controlled, adaptive phase II/III clinical study. The aim is to compare neoadjuvant chemotherapy of Docetaxel，Oxaliplatin combined with S-1(DOS) versus Oxaliplatin combined with S-1(SOX) in locally advanced gastric adenocarcinoma

DETAILED DESCRIPTION:
This trial is conducted in patients with locally advanced gastric adenocarcinoma. Eligible patients are randomized into two arms at 1:1 ratio to receive Docetaxel, Oxaliplatin combined with S-1(DOS) for 4 cycles or Oxaliplatin combined with S-1(SOX) for 3 cycles as neoadjuvant chemotherapy. All eligible patients will receive D2 gastrectomy if possible. Then, all eligible patients will also received DOS for 4 cycles or SOX for 3 cycles within 8 weeks after surgery. Study evaluation time is until death of patients or deadline set by the researchers.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory males or females with ages ≥ 18.
2. Karnofsky performance status ≥ 70%.
3. Histologically confirmed gastric adenocarcinoma including Lauren classification and validated overexpression of HER2.
4. cTNM should be diagnosed by enhanced CT/MRI (combined with endoscopic ultrasonography and diagnostic laparoscopic exploration) as cIII/IVa according to AJCC 8th classification.
5. Radical resection is possible before operation.
6. Research center and surgeons have the ability of conducting D2 lymphadenectomy (more than 15 lymph glands should be checked to ensure the quality of operation).
7. Physiological status and organ function are acceptable for major abdominal surgical operation.
8. Baseline blood routine and biochemical indexes of patients enrolled should meet criteria below: hemoglobin ≥ 90g/L, absolute neutrophil count ≥ 1.5×10⁹/L, platelet count ≥ 100×10⁹/L, aspartate or alanine aminotransferase ≤ 2.5 times the upper limit of normal (ULN), alkaline phosphatase ≤ 2.5 times the ULN, total serum bilirubin < 1.5 times the ULN, serum creatinine < 1 time ULN, Serum albumin ≥ 30g/L.
9. Left ventricular ejection fraction evaluated by echocardiac scanning ≥ 50%.
10. No severe comorbidity with less than 5 year survival.
11. Willing to receive the regimens in this study.
12. Sign written informed consent form before screening of study, and can withdraw in any time with no loss.
13. Agree to provide blood sample and histological specimen.

Exclusion Criteria：

1. Pregnancy or lactation women.
2. Woman of childbearing age was not tested in baseline pregnancy test or tested positve. Postmenopausal women with amenorrhea for at least 12 months are considered nonpregnancy.
3. Sexually active males or females refuse to practice contraception during the study.
4. With distant metastasis diagnosed by CT/EUS.
5. Underwent prior antitumor treatment including chemotherapy, radiotherapy or immunotherapy except steroid therapy.
6. Suffered from other malignant tumors in previous 5 years, with the exception of cured cutaneum carcinoma and cervical carcinoma in situ.
7. Patients with uncontrolled seizure, central nervous system disorder or psychiatric disease will be judged by researchers whether severity influences signing informed consent or compliance to take medicine.
8. Suffered from severe cardiovascular diseases such as symptomatic coronary heart disease, congestive heart failure ≥ II grade according to NYHA (New York Heart Association) standard, uncontrolled cardiac arrhythmia, cardiac infarction within 12 months prior to study enrollment.
9. Complicated by upper gastrointestinal obstruction or abnormal digestive function or malabsorption syndrome, which may affect the absorption of S-1.
10. Known peripheral nervous system disorder ≥ NCI CTC AE 1 grade with the exception of only disappearance of deep tendon reflex (DRT).
11. History of organ transplantation with immunosuppression therapy.
12. Complicated with severe uncontrolled concurrent infection or other severe uncontrolled concominant diseases, moderate or severe kidney injury (creatinine clearance rate ≤ 50 ml/min according to Cockcroft and Gault formula), or serum creatinine serum > the upper limit of normal (ULN)
13. Lack of dihydropyrimidine dehydrogenase (DPD).
14. Allergic reaction to platinum compounds or other agents used in this study.
15. Patients who have received study agents within 4 weeks (participating in other clinical trials).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The rate of pathologic complete response（pCR%） | 1 year
  Evaluation of pCR% of DOS regimen versus SOX regimen in locally advanced gastric adenocarcinoma

SECONDARY OUTCOMES:
Overall Survival : From date of enrollment until the date of death | 5 years
  Evaluation of the Overall Survival of DOS regimen versus SOX regimen in locally advanced gastric adenocarcinoma
Progression-free Survival：From date of enrollment until the date of first documented progression or second gastric cancer or death from any cause, whichever came first. | 3 years
  Evaluation of the Progression-free Survival of DOS regimen versus SOX regimen in locally advanced gastric adenocarcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, Professor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China